CLINICAL TRIAL: NCT04204889
Title: Trial of Oxaloacetate in Amyotrophic Lateral Sclerosis
Brief Title: Trial of Oxaloacetate in ALS
Acronym: TOALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Omar Jawdat (Other)
Collaborators: Terra Biological LLC (Industry)
Responsible Party: Sponsor-Investigator, Omar Jawdat, Principal Investigator, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOALS
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: ALS
MeSH Terms: interventions — Oxaloacetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oxaloacetate (Experimental): 3+3 dose escalating trial starting with 500mg twice daily orally and ending with 2500mg twice daily.
  Interventions: Drug: Oxaloacetic Acid

INTERVENTIONS:
Drug: Oxaloacetic Acid — The first 3 patients will receive 500 mg twice daily, and subsequent cohorts will increase by 500 mg per dose to a maximum of 2500 mg twice daily.
  Other Names: Oxaloacetate

SUMMARY:
The purpose of this study is to determine the safety and the maximal tolerated dose of Oxaloacetate (OAA) in patients with Amyotrophic Lateral Sclerosis (ALS).

DETAILED DESCRIPTION:
Overview This is a safety and dose finding study looking at Oxaloacetate (OAA) in patients with Amyotrophic Lateral Sclerosis (ALS). This study will aim to determine the maximal dose that a subject can tolerate. The investigators will also learn how OAA affects mitochondria in subjects with ALS. This is a 28-day study in which the investigators will attempt to enroll approximately 24 participants. There is no placebo control.

Specific Aims (Hypothesis and Objectives)

The overall goal of this proposal is to determine if reducing mitochondrial stress is a viable treatment strategy for ALS. This study will determine the maximal tolerated dose of OAA and whether OAA improves biomarkers of mitochondrial stress. ALS is a progressive fatal neurodegenerative disorder caused by loss of motor neurons in the brain and spinal cord. Despite multiple clinical trials and advances in understanding of the pathogenesis of ALS, riluzole and edaravone, the only Food and Drug Administration (FDA) approved ALS drugs, the former only extends life by a few months, and the latter possibly slows down functional decline. Hence there is a clear need for new treatments for ALS.

While the exact underlying cause of this motor neuron degeneration remains uncertain, candidate mechanisms include glutamate excitotoxicity, free radical-mediated oxidative cytotoxicity, neuroinflammation, mitochondrial dysfunction, autoimmune processes, protein aggregation, and cytoskeletal abnormalities. Mitochondrial dysfunction in particular may play a critical role in ALS neurodegeneration, an observation supported by both human and animal model studies. The characteristic pathological ALS finding of cytoplasmic inclusions (Bunina bodies) in motor neuron cell bodies may represent mitochondria-containing autophagic vacuoles. Functional studies of ALS mitochondria were also reported: calcium levels in motor neuron synaptic terminals of ALS subjects were found to be elevated despite increased numbers of local mitochondria, suggesting a defect of mitochondrial calcium sequestration; increased complex I activity was seen with familial ALS; and reduced cytochrome oxidase activity was shown in sporadic ALS patients. In mutant SOD mouse model, evidence of mitochondrial dysfunction appears before motor neuron degeneration. Similar observations have been noted in human sporadic ALS tissue. In humans with pathogenic mutations in TARDBP and C9ORF72, mitochondrial functionality is abnormal in peripheral fibroblasts. The dexpramipexole trial in ALS, while negative, is based on the mitochondrial ALS pathogenesis theory. The investigators performed an open label study of rasagiline in ALS and demonstrated target engagement of several blood mitochondrial biomarkers. KUMC completed an 80 patient randomized controlled trial of rasagiline in ALS and again measured mitochondrial biomarkers.

Rationale: Human and animal studies suggest targeting mitochondrial dysfunction may be an important approach to slow disease progression in ALS. Mitochondrial dysfunction can be seen in both in vitro and in vivo experimental ALS models, may explain the characteristic Bunina bodies, a key ALS pathological hallmark, and mitochondrial abnormalities are found in patient autopsies. In cell models of mitochondrial dysfunction, OAA has been shown to be cytoprotective. In addition, there is evidence that OAA, in preclinical studies in Alzheimer disease, reduces neuroinflammation, another possible ALS pathological pathway. A phase 2 trial of OAA in in Alzheimer Disease is currently being conducted at KUMC but at a lower dose than is proposed in this ALS study. The investigator is interested in OAA as a potential therapeutic agent in ALS as it crosses the blood brain barrier, accesses motor neurons, activates mitochondrial bioenergetics, increases respiratory capacity, and increases glycolysis capacity. Preliminary data of OAA in an ALS mouse model at KUMC increased muscle strength compared to untreated animals.

Hypothesis: OAA will be neuroprotective in ALS by reducing mitochondrial stress. This trial will determine whether OAA is tolerable and whether it engages mitochondrial targets in ALS patients. The result of this trial will lead to a larger phase II trial to further assess safety and to begin to study efficacy in slowing the disease process. This short 28 day study is too brief to study efficacy.

Specific Aim 1: To determine safety and the maximal tolerated dose of OAA in patients with ALS. To achieve this aim, the investigator will conduct a prospective 3 + 3 dose escalating clinical trial in up to 24 clinically definite, probable, or laboratory supported probable ALS patients.

Sub-aim 1: The investigator will determine the pharmacokinetic profile of OAA in ALS patients. The investigator will evaluate OAA drug levels in a pre-dose sample, 1 hour and 4 hours after dosing.

Specific Aim 2: To determine OAA target engagement. The investigator will evaluate a panel of mitochondrial biomarkers, platelet TDP-43 levels and MR spectroscopy of brain glutathione, at baseline then at the end of treatment and compare biomarker levels to dose, to evaluate possible dose-response relationship in our biomarkers.

Future Aim: The goal is to use the results from this study to conduct a larger prospective placebo controlled trial to determine if OAA is well tolerated and slows disease progression in ALS using the maximal tolerated dose that will be determined during this current study

.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis by a study investigator of laboratory-supported probable, probable, or definite ALS, according to the modified El Escorial criteria[1]
* Vital capacity (VC) greater or equal to 50% of predicted
* Diagnosis with ALS within 3 years prior to enrollment
* If patients are taking riluzole for ALS, they must be on a stable dose for at least thirty days prior to the baseline visit
* Women of childbearing age must use protection against pregnancy.

Exclusion Criteria:

* Requirement for tracheotomy ventilation or non-invasive ventilation for > 23 hours per day
* Diagnosis of other neurodegenerative diseases (e.g., Parkinson disease, Alzheimer disease)
* Clinically significant history of unstable medical illness (e.g., unstable angina, advanced cancer) over the last 30 days
* Current pregnancy or lactation
* Limited mental capacity such that the patient cannot provide written informed consent or comply with evaluation procedures
* Receipt of any investigational drug within the past 30 days from enrollment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | Day 28
  Defined as any serious adverse event related to OAA requiring hospitalization, or any AE related to OAA requiring stopping the medication, including a two fold increase in AST and/or LAT and /or a 1.5 times increase in creatinine level.

SECONDARY OUTCOMES:
Pharmacokinetic testing | Day 28
  OAA Levels
Mitochondrial Biomarkers | Day 28
  Annexin V/Mitotracker in lymphocytes: assess modification of apoptosis/mitochondrial number. TMRE: Mitochondrial membrane potential. MitoSox: Mitochondrial superoxide. Glutamate-plasma: OAA specific biomarker.
Platelet Biomarker | Day 28
  The levels of Serum TDP43
MR spectroscopy | Day 28
  MR spectroscopy of brain glutathione

CONTACTS AND LOCATIONS:
Overall Officials: Omar Jawdat, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States